CLINICAL TRIAL: NCT04798261
Title: STRIKE-PE: A Prospective, Multicenter Study of the Indigo™ Aspiration System Seeking to Evaluate the Long-Term Safety and Outcomes of Treating Pulmonary Embolism
Brief Title: Study of the Long-Term Safety and Outcomes of Treating Pulmonary Embolism With the Indigo Aspiration System
Status: Recruiting | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18135
Record Dates: First submitted 2021-02-26; First posted 2021-03-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with acute pulmonary embolism
  Interventions: Device: Indigo Aspiration System

INTERVENTIONS:
Device: Indigo Aspiration System — Indigo Aspiration System

SUMMARY:
The objective of this study is to evaluate real world long-term functional outcomes, safety and performance of the Indigo Aspiration System for the treatment of pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs and symptoms consistent with acute PE with duration of 14 days or less
2. RV/LV ratio ≥ 0.9 assessed by diagnostic computed tomographic angiography (CTA) or echocardiogram
3. Frontline endovascular treatment with the Indigo Aspiration System per IFU
4. Patient is ≥ 18 years of age
5. Informed consent obtained per Institutional Review Board/Ethics Committee requirements

Exclusion Criteria:

1. Contraindication to systemic or therapeutic doses of anticoagulants (e.g. heparin)
2. Stage IV (metastatic) cancer, active lung cancer or previous history of surgery in the affected lung(s) or chest radiation
3. Known serious, uncontrolled sensitivity to radiographic agents
4. Life expectancy < 180 days
5. Patients on ECMO
6. Pregnant patients
7. Current participation in another investigational drug or device study that may confound the results of this study. Studies requiring extended follow-up for products that were investigational but have since become commercially available are not considered investigational studies
8. Other medical, social, or psychological conditions that, in the opinion of the Investigator, precludes the patient from appropriate consent, could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Safety: Composite of major adverse events | 48 hours
  A composite of device-related death, major bleeding, device-related clinical deterioration, device-related pulmonary vascular injury and device-related cardiac injury
Performance: Change in RV/LV Ratio | 48 hours post-procedure
  Change in RV/LV Ratio (matched imaging pairs CTA or echocardiogram, as available)

SECONDARY OUTCOMES:
Quality of Life assessed via PEmb-QoL | 90 days post-procedure
  Self-assessment of PE related complaints and daily living limitations (including work and social)
Quality of Life assessed via EQ-5D-5L | 90 days post-procedure
  Self-assessment of activities of daily living
Functional outcome assessed NYHA | 90 days post-procedure
  Physician assessment of heart failure symptoms and activity level
Functional outcome assessed via 6MWT | 90 days post-procedure
  Walking distance over a 6 minute period to assess functional capacity
Perceived dyspnea assessed via Borg Scale | 90 days post-procedure
  Category rating scale to measure perceived dyspnea
Incidence of device related SAE(s) | 365 days
Any-cause mortality | Within 30 days
Symptomatic PE recurrence | Within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: John Moriarty, MD, Principal Investigator — University of California, Los Angeles; Ido Weinberg, MD, Principal Investigator — Massachusetts General Hospital
Locations (71):
- United States (54):
  - Long Beach Medical Center, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - Christiana Care Hospital, Newark, Delaware
  - Manatee Memorial Hospital, Bradenton, Florida
  - Blake Medical Center/Nova Clinical Research, Brandenton, Florida
  - Delray Medical Center, Inc., Delray Beach, Florida
  - University of Florida Shands Hospital, Gainesville, Florida
  - Radiology and Imaging Specialists, Lakeland, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Baptist Health Miami Cardiac and Vascular Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - HCA Florida Northside Hospital, Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Joseph Hospital - BayCare, Tampa, Florida
  - University Hospital Augusta, Augusta, Georgia
  - Memorial Hospital Belleville, Belleville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - KUMC, Kansas City, Kansas
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - Ascension St. John Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Hospital South, St Louis, Missouri
  - Cooper Health System, Camden, New Jersey
  - Lovelace Health System, Albuquerque, New Mexico
  - Bellevue Hospital Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - St. Francis Hospital and Heart Center, Roslyn, New York
  - Staten Island University Hospital, Staten Island, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - TriHealth Good Samaritan Hospital, Cincinnati, Ohio
  - Mount Carmel East, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - UPMC Harrisburg, Harrisburg, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Methodist Hospital Metropolitan, San Antonio, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Christus Mother Frances Hospital, Tyler, Texas
  - Sentara Norfolk General, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Flinders Medical Centre, Bedford Park, South Australia, Australia
- Hospital Santa Lucia Sul, Brasília, Brazil
- Germany (2):
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - GRN-Klinik Weinheim, Weinheim
- Italy (2):
  - Ospedale Misericordia, Grosseto
  - Ospedale San Giovanni Bosco, Torino
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Poland (4):
  - Krakowski Szpital Specjalistyczny św. Jana Pawła II, Krakow
  - Europejskie Centrum Zdrowia Otwock, Otwock
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
- Hospital de Santa Cruz, Carnaxide, Portugal
- Spain (2):
  - Hospital Universitario Virgen de la Nieves, Granada
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- United Kingdom (3):
  - Royal Sussex County Hospital, Brighton, Sussex
  - University Hospital of Wales, Cardiff, Wales
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moriarty JM, Schiro BJ, Dohad SY, Tamaddon H, Davis HC, Shavelle DM, Chrysant GS, Iliadis EA, Dexter DJ 2nd, Ciampi Dopazo JJ, Holden A, West FM, Keeling B, Sharp ASP, Weinberg I. Periprocedural Results and Right Ventricular Outcomes of Computer Assisted Vacuum Thrombectomy Treatment of Acute Pulmonary Embolism: Interim Analysis of 300 Patients From the STRIKE-PE Study. J Am Heart Assoc. 2025 Sep 2;14(17):e039975. doi: 10.1161/JAHA.124.039975. Epub 2025 Aug 29. PMID 40878986